CLINICAL TRIAL: NCT04151901
Title: Sex-specific Determinants of Early-phase Recovery From Skeletal Muscle Disuse
Acronym: MAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: HSC20230594H; R01AG064386 (NIH)
Record Dates: First submitted 2019-10-09; First posted 2019-11-05 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Atrophy of Muscle Due to Disuse; Rehabilitation
MeSH Terms: conditions — Muscular Disorders, Atrophic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Male Rehabilitation (M-REHAB) (Experimental): Disuse + resistance exercise rehabilitation
  Interventions: Other: Resistance Exercise Rehabilitation
- Male Control (M-CON) (Experimental): Disuse + ambulatory control rehabilitation
  Interventions: Other: Walking-based rehabilitation
- Female Rehabilitation (F-REHAB) (Experimental): Disuse + resistance exercise rehabilitation
  Interventions: Other: Resistance Exercise Rehabilitation
- Female Control (F-CON) (Experimental): Disuse + ambulatory control rehabilitation
  Interventions: Other: Walking-based rehabilitation

INTERVENTIONS:
Other: Resistance Exercise Rehabilitation — Following disuse, the REHAB groups (M-REHAB, F-REHAB) will complete monitored resistance exercise rehabilitation sessions using an isokinetic dynamometer at a similar relative load at each rehab visit.
  Arms: Female Rehabilitation (F-REHAB); Male Rehabilitation (M-REHAB)
Other: Walking-based rehabilitation — Following disuse, the CON groups (M-CON, F-CON) will complete 30 minutes of monitored walking at a moderate intensity at each rehab visit.
  Arms: Female Control (F-CON); Male Control (M-CON)

SUMMARY:
This project is a 2-phase, randomized clinical trial that includes 7 days of unilateral leg disuse (Phase 1), immediately followed by 1 week of bilateral leg rehabilitation (Phase 2). The investigators will recruit cohorts of healthy middle-aged men and women to address their aims:

* Demonstrate the sex-specific effects of skeletal muscle disuse (Phase 1)
* Identify key molecular determinates of susceptibility of skeletal muscle atrophy (Phase 1)
* Map the early, sex-specific molecular time-course of rehabilitation (Phase 2)
* Determine if disused and healthy muscle respond similarly to exercise (Phase 2)

Healthy, middle-age men and post-menopausal women (50-65 years) will be recruited from the greater Houston/Galveston area. This under-represented research demographic demonstrate few negative metabolic or phenotypic signs of advanced age, but are at increased risk of being hospitalized and experiencing accelerated loss of lean mass and muscle function that parallels a much older population.

The goal of this study is to characterize phenotypic and molecular skeletal muscle changes in middle-aged men and women during critical periods of disuse and rehabilitation and ultimately direct the development of targeted and effective prevention and treatment strategies.

DETAILED DESCRIPTION:
The negative health consequences of muscular disuse in aging populations are unequivocal. While descriptive, outcome data on disuse and recovery are abundant, key knowledge gaps limit researcher's ability to implement evidence-based, rehabilitation strategies. Limiters include: i) an inability to identify individuals most susceptible to disuse, ii) insufficient information to differentiate between, and respond to, disuse atrophy in men and women, iii) limited insight into the mechanisms driving adaptation to early rehabilitative exercise, and iv) the assumption that disused and healthy skeletal muscle will have a similar, positive response to resistance exercise. The investigators will complete a 2-phase, randomized clinical trial. The protocol includes 7-days of unilateral leg disuse (ULD; Phase 1), immediately followed by 1 week of bilateral leg rehabilitation (Phase 2). Healthy, middle-aged men (n=40) and (post-menopausal) women (n=40), (50-65 y) will be recruited; a neglected research demographic who present with a largely youthful phenotype, but are at risk of accelerated disuse atrophy.

This project will provide a highly powered, detailed phenotypic characterization of the continuum of adults most and least susceptible to muscular disuse. Clinical outcomes will be supported by RNA deep sequencing and pathway analysis to establish a platform that: i) improves scientists' ability to identify higher-risk individuals and ii) provides insight into time-sensitive, sex-specific and effective rehabilitation strategies. Findings and reposed molecular data from this study, may help identify future therapeutic targets and serve as an uncomplicated/comorbidity-free baseline for clinical trials in populations experiencing disuse atrophy.

ELIGIBILITY:
Inclusion Criteria:

1. All races and ethnic backgrounds
2. Men and women, age 50-65 years
3. Generally healthy (see exclusion criteria)
4. Able and willing to provide informed consent
5. Ability to speak and read English
6. Post-menopausal women (no menses within the last 12 months)
7. Body mass index: 18.5-35 kg/m2 or BMI>35 if thigh adiposity does not impair muscle biopsy

Exclusion Criteria:

1. Compromised musculoskeletal function that precludes safe participation or use of crutches
2. Pre-menopausal women
3. Hypogonadal men (testosterone <300 ng/dL)
4. Women taking hormone replacement therapy (HRT)
5. Sarcopenia (European Working Group on Sarcopenia in Older People, EWGSOP102)
6. Clinically significant heart disease (e.g. New York Heart Classification greater than grade II; ischemia)
7. Peripheral vascular disease
8. History of claudication
9. Pulmonary disease
10. History of systemic or pulmonary embolus
11. Uncontrolled blood pressure (systolic BP>170, diastolic BP>95 mmHg)
12. Impaired renal function (creatinine >1.5 mg/dl)
13. Anemia (hematocrit <33)
14. Untreated thyroid disease (abnormal TSH)
15. A recent history (<12 months) of GI bleed
16. Diabetes mellitus or other untreated endocrine or metabolic disease
17. Electrolyte abnormalities
18. Any history of stroke, hypo- or hyper-coagulation disorders
19. Employment requiring long (>1 h) uninterrupted period of standing
20. Inability to meet study travel requirements (e.g. manual geared car)
21. Recent history of balance issues or falls.
22. Recent (3 years) treated cancer other than basal cell carcinoma
23. Systemic steroids, anabolic steroids, growth hormone or immunosuppressant use within 12 months
24. Recent (2 months) adherence to a weight-loss or weight-gain diet
25. Weight change of 5% or more in previous 6 months
26. Body mass index >30 or excess body fat that compromises muscle biopsy collection
27. Acute infectious disease or chronic infection
28. Alcohol or drug abuse
29. Any other condition or event considered exclusionary by study physician

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-08-27 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Quantitative RNA-sequencing | Study day 1 (before starting leg disuse)
  RNA deep sequence analysis on muscle tissue taken from a muscle biopsy to measure transcriptome
Quantitative RNA-sequencing | Study day 7 (after finishing leg disuse)
  RNA deep sequence analysis on muscle tissue taken from a muscle biopsy to measure transcriptome
Quantitative RNA-sequencing | Study day 7 (after 1 bout of rehabilitation)
  RNA deep sequence analysis on muscle tissue taken from a muscle biopsy to measure transcriptome
Quantitative RNA-sequencing | Study day 9 (after 2 bouts of rehabilitation)
  RNA deep sequence analysis on muscle tissue taken from a muscle biopsy to measure transcriptome
Quantitative RNA-sequencing | Study Day 11 (after 3 bouts of rehabilitation)
  RNA deep sequence analysis on muscle tissue taken from a muscle biopsy to measure transcriptome
Quantitative RNA-sequencing | Study Day 21 (after finishing 7 bouts of rehabilitation)
  RNA deep sequence analysis on muscle tissue taken from a muscle biopsy to measure transcriptome
Muscle function | Study day 1 (before starting leg disuse)
  Each leg will be individually tested on an isokinetic dynamometer to determine muscle strength (peak torque)
Muscle function | Study day 7 (after 1 bout of rehabilitation)
  Each leg will be individually tested on an isokinetic dynamometer to determine muscle strength (peak torque)
Muscle function | Study day 9 (after 2 bouts of rehabilitation)
  Each leg will be individually tested on an isokinetic dynamometer to determine muscle strength (peak torque)
Muscle function | Study Day 11 (after 3 bouts of rehabilitation)
  Each leg will be individually tested on an isokinetic dynamometer to determine muscle strength (peak torque)
Muscle function | Study Day 21 (after finishing 7 bouts of rehabilitation)
  Each leg will be individually tested on an isokinetic dynamometer to determine muscle strength (peak torque)
Body (leg) composition | Study day 1 (before starting leg disuse)
  Leg lean mass will be assessed via segmental dual energy x-ray absorptiometry
Body (leg) composition | Study day 7 (after finishing leg disuse)
  Leg lean mass will be assessed via segmental dual energy x-ray absorptiometry
Body (leg) composition | Study day 9 (after 2 bouts of rehabilitation)
  Leg lean mass will be assessed via segmental dual energy x-ray absorptiometry
Body (leg) composition | Study Day 11 (after 3 bouts of rehabilitation)
  Leg lean mass will be assessed via segmental dual energy x-ray absorptiometry
Body (leg) composition | Study Day 21 (after finishing 7 bouts of rehabilitation)
  Leg lean mass will be assessed via segmental dual energy x-ray absorptiometry

SECONDARY OUTCOMES:
Muscle fiber cross sectional area | Study day 1 (before starting leg disuse)
  Muscle biopsy samples will be evaluated for muscle fiber cross sectional area
Muscle fiber cross sectional area | Study day 7 (after finishing leg disuse)
  Muscle biopsy samples will be evaluated for muscle fiber cross sectional area
Muscle fiber cross sectional area | Study day 9 (after 2 bouts of rehabilitation)
  Muscle biopsy samples will be evaluated for muscle fiber cross sectional area
Muscle fiber cross sectional area | Study Day 11 (after 3 bouts of rehabilitation)
  Muscle biopsy samples will be evaluated for muscle fiber cross sectional area
Muscle fiber cross sectional area | Study Day 21 (after finishing 7 bouts of rehabilitation)
  Muscle biopsy samples will be evaluated for muscle fiber cross sectional area
Muscle fiber type | Study day 1 (before starting leg disuse)
  Muscle biopsy samples will be evaluated for muscle fiber type distribution
Muscle fiber type | Study day 7 (after finishing leg disuse)
  Muscle biopsy samples will be evaluated for muscle fiber type distribution
Muscle fiber type | Study day 9 (after 2 bouts of rehabilitation)
  Muscle biopsy samples will be evaluated for muscle fiber type distribution
Muscle fiber type | Study Day 11 (after 3 bouts of rehabilitation)
  Muscle biopsy samples will be evaluated for muscle fiber type distribution
Muscle fiber type | Study Day 21 (after finishing 7 bouts of rehabilitation)
  Muscle biopsy samples will be evaluated for muscle fiber type distribution
Diet recall | Familiarization session (~1 week before starting leg disuse)
  A multi-pass 24-hour dietary recall using the Automated Self Assessment 24-h dietary assessment tool to determine habitual food intake
Diet recall | Study day 11 (after two bouts of rehabilitation)
  A multi-pass 24-hour dietary recall using the Automated Self Assessment 24-h dietary assessment tool to determine habitual food intake
Physical activity | Study Days -7 to Day 0 (1 week prior to starting leg disuse)
  Accelerometers will placed on the waist and ankle to measure physical activity
Physical activity | Study Days 1-6 (1 week of disuse)
  Accelerometers will placed on the waist and ankle to measure physical activity
Physical activity | Study Days 7-21 (2 weeks of rehabilitation)
  Accelerometers will placed on the waist and ankle to measure physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Blake Rasmussen, PhD, Principal Investigator — University of Texas Health Science Center as San Antonio
Locations (2):
- United States (2):
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
All collected de-identified Individual Participant Data (IPD) that underlie results in a publication. Biological samples will not be available to other/outside investigators, but may be used by the research team for future related assays and experiments.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be shared at study completion as summary results on ClinicalTrials.gov and after review and publication in a peer-reviewed journal.